CLINICAL TRIAL: NCT02752269
Title: Early Detection of Pulmonary- and Pulmonary Vascular Disease in Patients Suffering From Sjögren Syndrome
Brief Title: Early Detection of Pulmonary- and Pulmonary Vascular Disease in Sjögren Syndrome
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 26-446 ex 13/14
Record Dates: First submitted 2015-11-24; First posted 2016-04-26 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Sjögren Syndrome; Pulmonary Hypertension
MeSH Terms: conditions — Sjogren's Syndrome; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
According to the literature available pulmonary hypertension is present in 12 to 23% of patients suffering from Sjögren Syndrome. However epidemiological data are based on non-invasive measurements using echocardiography. Furthermore, no data are available regarding exercise hemodynamics in those patients.

This study investigates pulmonary hemodynamics at rest and during exercise in patients suffering from primary and secondary Sjögren Syndrome. Patients under suspicion for pulmonary hypertension (PH) will be offered further investigations including right heart catheterization.

DETAILED DESCRIPTION:
Patients with primary and secondary Sjögren Syndrome will be investigated using echocardiography, exercise echocardiography, pulmonary function testing, laboratory testing, electrocardiogram and 6 minute walking test. Those patients under clinical suspicion for pulmonary hypertension will be offered further investigations including right heart catheterization to rule out or verify the diagnosis of manifest pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* informed Consent
* diagnosis of Sjögren Syndrome
* age: 18 - 90 yrs

Exclusion Criteria:

* uncontrolled systemic hypertension (at rest >150 mmHg systolic or 95 mmHg diastolic)
* relevant systolic (EF<50%) or diastolic (>Grade 1) left ventricular dysfunction
* uncontrolled ventricular arrhythmias
* uncontrolled supraventricular bradycardia or tachycardia
* myocardial infarction within the last 12 months
* pulmonary embolism within the last 6 months
* larger surgical interventions within the last 12 months
* musculoskeletal or vascular disease, that may affect ergometric investigations
* pregnancy (anamnesis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary Sjögren Syndrome.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-10; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
prevalence of pulmonary hypertension in Sjögren syndrome | 2 hours
  % of patients with mean pulmonary arterial pressure > 25 mmHg

SECONDARY OUTCOMES:
forced vital capacity | 2 hours
  % predicted
systolic pulmonary arterial pressure at 50 Watts | 2 hours
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — MUG
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No